CLINICAL TRIAL: NCT01112007
Title: Searching for Accomplices in the Transgression of Insulin Resistance in Prehypertension: Aldosterone?
Brief Title: Accomplices of Insulin Resistance in Prehypertension: Aldosterone?
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Attending physician, Taipei Veterans General Hospital, Taiwan
Other Study IDs: V99C1-153
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Hypertension; Insulin Resistance
Keywords: Insulin Resistance; Hypertension; Blood pressure; Aldosterone; Renin
MeSH Terms: conditions — Hypertension; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- prehypertension: Subjects with prehypertension, that is, individuals with systolic blood pressure in the range of 120-139 mmHg or diastolic BP between 80-89 mmHg.

SUMMARY:
The purposes of the study are to evaluate the relative contributions of insulin resistance and renin-angiotensin-aldosterone system to blood pressure (BP) in subjects with prehypertension. This is a cross-sectional study. Anthropometric and BP measurements will be performed in 50 prehypertensive subjects. The subjects will receive a 75-g oral glucose tolerance test and a postural stimulation test for the measurements of insulin resistance, plasma rennin concentration and aldosterone level. Log (ISI0,120), an insulin sensitivity index from the oral glucose tolerance test, will be calculated. Statistical analyses will be performed to compare the degree to which aldosterone and Log (ISI0,120) predicted systolic and diastolic BP in these prehypertensive subjects.

DETAILED DESCRIPTION:
Background: Prehypertension, a new category of blood pressure (BP) classification introduced by The Seven Report of the Joint National Commission (JNC-7) on High BP for individuals with systolic BP in the range of 120-139 mmHg or diastolic BP between 80-89 mmHg, is a strong predictor for the development of hypertension. Insulin resistance (IR) is reported to be associated with prehypertension. Activation of the renin-angiotensin-aldosterone (RAA) system is a major player in IR and elevation of high BP.

Aim: The purposes of the study are to evaluate the interactions of IR-RAA and their relative contributions to BP in subjects with prehypertension.

Design: This is a cross-sectional study. Methods: Anthropometric and BP measurements will be performed in 50 prehypertensive subjects. The subjects will receive a 75-g oral glucose tolerance test (OGTT) and a postural stimulation test for the measurements of IR, plasma rennin concentration (PRC) and aldosterone level. The study participants will be divided into three subgroups by tertiles of Log (ISI0,120), an insulin sensitivity index from the OGTT. Analysis of variance (ANOVA) will be applied to compare the differences in clinical characteristics among the three groups. Univariate analyses of general linear models will be used to compare the differences in PRC, aldosterone, and aldosterone/rennin ratio (ARR) in postural stimulation tests among the three subgroups, showing effects of confounding variables including age, sex, BMI and physical inactivity scores. Repeated-measures ANOVA will be used to assess the differences in post-challenge PRC, aldosterone, and ARR responses in the OGTT with or without adjustments of the above covariates. Pearson and partial correlation procedures will be used to test the correlations of PRC, aldosterone, ARR with insulin sensitivity and BP. Multiple linear regression models will be used in an attempt to compare the degree to which aldosterone (or ARR) and Log (ISI0,120) predicted systolic and diastolic BP in these prehypertensive subjects.

Expected results and contributions: We hope the study can explore the contribution of the IR-RAA interactions to BP in subjects with prehypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 20 - 70 years old.
2. Subjects with prehypertension,; that is, individuals with systolic blood pressure (BP) in the range of 120-139 mmHg or diastolic BP between 80-89 mmHg.
3. Willing to participate by signing an informed consent.
4. Willing to undergo two clinical tests at two separate visits.

Exclusion Criteria:

1. Patients with known history of type 2 diabetes or fasting plasma glucose greater than 126 mg/dL.
2. Patients with known history of hypertension.
3. History of major renal, liver, heart, blood and neurological disease.
4. History of alcoholism or drug abuse.
5. Women who are pregnant.
6. Current or concomitant illness that would interfere with the subject's ability to perform the study or that would confound the study results, judged by the investigation physicians.
7. Any concomitant BP-lowering, anti-lipid, and glucose-modification agents within 2 weeks of the study, and oral contraceptives and estrogen therapy within 8 weeks of the study.
8. Difficult venous access.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with prehypertension, that is, individuals with systolic blood pressure (BP) in the range of 120-139 mmHg or diastolic BP between 80-89 mmHg.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Renin and aldosterone responses in postural stimulation tests | 2 weeks
  The differences in renin and aldosterone responses in postural stimulation tests among the three subgroups, showing effects of confounding variables including age, sex, body mass index (BMI) and physical inactivity scores

SECONDARY OUTCOMES:
The differences in post-challenge renin and aldosterone responses in the oral glucose tolerance | 2 weeks
  Repeated-measures analysis of variance (ANOVA) will be used to assess the differences in post-challenge renin and aldosterone responses in the oral glucose tolerance test with or without adjustments.
Correlations of renin and aldosterone with insulin sensitivity | 2 weeks
  Pearson and partial correlation procedures will be used to test the correlations of renin and aldosterone with insulin sensitivity.
Correlations of renin and aldosterone with blood pressure | 2 weeks
  Pearson and partial correlation procedures will be used to test the correlations of renin and aldosterone with blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Min Hwu, MD, Principal Investigator — Section of Endocrinology and Metabolism, Department of Medicine, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan